CLINICAL TRIAL: NCT05730530
Title: Nutrition Education Intervention to Improve Fruit and Vegetable Consumption in Preschoolers
Brief Title: Fruit and Vegetable Intake in Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Sibylle Kranz, PhD, RDN, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBS 5304
Record Dates: First submitted 2023-02-01; First posted 2023-02-16 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Children, Only; Nutrition, Healthy
Keywords: Preschool; Fruits and vegetables; Nutrition education; Behavior change theory

STUDY DESIGN:
Intervention Model Description: Group-randomized trial with individual-level outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Classroom assigned to receive the 6-week long nutrition education curriculum
  Interventions: Behavioral: Nutrition education curriculum
- Control (No Intervention): Classroom assigned to receive no intervention

INTERVENTIONS:
Behavioral: Nutrition education curriculum — This intervention consists of a 6-week-long nutrition education curriculum aimed at improving fruit and vegetable acceptance and consumption. Sessions will occur within the classroom 3 times per week for 6 weeks. Each week, the sessions will consist of 2 days of teaching activities and 1 day of taste-test activities designed for children to guess various common fruits and vegetables, assemble recipes including 2-4 different fruits and vegetables, and then taste the foods. These activities will be conducted in a full-classroom group setting.
  Arms: Intervention

SUMMARY:
The goal of this randomized controlled trial is to examine fruit and vegetable consumption in preschoolers following a nutrition education curriculum. The main questions it aims to answer is:

1. Is this intervention consisting of nutrition education and taste-test activities able to improve fruit and vegetable consumption in preschoolers during their usual lunch meal?
2. Is the improvement of fruit and vegetable consumption sustained for at least 6 weeks after completion of the intervention?

Participants in the intervention classroom will partake in 3 nutrition education sessions per week during the 6-week-long curriculum. Researchers will compare this to changes in fruit and vegetable intake of the children in the control classroom, who will undergo identical measurements, but will not participate in the curriculum.

DETAILED DESCRIPTION:
Fruit and vegetable consumption in preschoolers in the United States is very low, with the majority of children not meeting the national recommendations. However, there is a lack of data indicating effective strategies to increase preschooler's fruit and vegetable intake and whether socio-demographic and eating behavior-related child characteristics (child eating behavior and relationship with food) may predict fruit and vegetable consumption in preschoolers as well as their response to the intervention. This information is important for researchers because it may allow for more effective development of future interventions that consider these potential external influences. There is also a lack of evidence-based interventions that are based on theoretical behavior change frameworks and the associated behavior change techniques. Furthermore, studies lack a long enough follow-up to measure whether any possibly observed behavior change (more fruits and vegetables consumed) in the preschoolers is maintained following the cessation of the intervention.

While fruit and vegetable consumption is associated with lower blood pressure in adults, little is known about this relationship in children. This will be examined in our study to determine if there is an association between blood pressure and fruit and vegetable intake at baseline and whether this association changes following the intervention.

To control for differences in energy needs, it is important to control for children's BMI-for-age percentile, which is calculated using their age, height, and weight. This is necessary because children who have higher BMI percentiles typically require more total energy consumption, which may influence fruit and vegetable consumption. Additionally, previous studies have observed that children with greater BMI percentile are less likely to eat adequate amounts of fruits and vegetables. However, this has not been measured in an interventional manner, and therefore it is unknown whether these associations are omnipotent, and whether they remain following a fruit and vegetable intervention. Therefore, our study will examine these relationships in a small sample of preschoolers to either support or contradict these previous observations.

In addition to measuring fruit and vegetable intake, it is also important to measure physical activity levels as a control variable for total energy requirements, as changes in physical activity levels may confound changes in dietary intake, including intake of fruits and vegetables. This is especially true of interventions that span different seasons (ie. winter and spring), as these may also influence physical activity levels and, subsequently, energy requirements. Secondarily, previous research has established an association between fruit and vegetable intake and both physical activity levels and screen time in children and adults. However, no studies have explored this relationship in preschool-aged children. Additionally, the evidence of the relationship between these two variables is limited to cross-sectional data; it is unknown whether an increase in one would influence the other. We plan to examine this in a small sample of preschoolers in an interventional setting.

Therefore, the purpose of this research is to determine whether such an intervention is able to increase and maintain fruit and vegetable intake during lunch in a sample of preschoolers, controlling for age, BMI percentile, and activity level. Additional aims are 1) to explore the relationship between fruit and vegetable intake and blood pressure, 2) examine the relationship between FV intake and physical activity levels in this sample of preschoolers, and 3) examine how BMI-percentile and socio-demographic and child- and parent-related eating-related characteristics are associated with fruit and vegetable intake. We plan to publish our findings in a scientific journal to contribute to the advancement of knowledge regarding interventions to improve fruit and vegetable intake in preschoolers, as information is evidently needed in this topic.

ELIGIBILITY:
Inclusion Criteria:

* Typically-developing children with no food allergies and not taking medication

Exclusion Criteria:

* Food Allergies
* Taking medications
* Developmental delays

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Fruit and vegetable intake post-intervention | Change in fruit and vegetable intake from baseline (week 0) to post-intervention (week 7)
  Fruits and vegetables consumed during a typical lunch meal, measured using plate-waste weighing method, which involves subtracting the grams of food leftover from the grams of food served to estimate the grams of food consumed. All weighing of the foods will be done in the Diet and Nutrition Lab before and after going to the childcare center. This will be measured on three consecutive days during each of the measurement weeks below.
Fruit and vegetable intake at follow-up | Change in fruit and vegetable intake from baseline (week 0) to follow-up (week 14)
  Fruits and vegetables consumed during a typical lunch meal, measured using plate-waste weighing method, which involves subtracting the grams of food leftover from the grams of food served to estimate the grams of food consumed. All weighing of the foods will be done in the Diet and Nutrition Lab before and after going to the childcare center. This will be measured on three consecutive days during each of the measurement weeks below.
Skin carotenoid levels post-intervention | Change in fruit and vegetable intake from baseline (week 0) to post-intervention (week 7)
  Children's fruit and vegetable intake will be confirmed using a measure of skin carotenoid levels. This will be measured using a VeggieMeter device, which utilizes non-invasive reflection spectroscopy to estimate the amount of dietary carotenoids deposited into the skin. Children will be asked to wash their hands and then place their right pointer finger on a small lens for approximately 15 seconds. This will be measured immediately following the 3 measured lunch meals at the 3 time points.
Skin carotenoid levels at follow-up | Change in fruit and vegetable intake from baseline (week 0) to follow-up (week 14)
  Children's fruit and vegetable intake will be confirmed using a measure of skin carotenoid levels. This will be measured using a VeggieMeter device, which utilizes non-invasive reflection spectroscopy to estimate the amount of dietary carotenoids deposited into the skin. Children will be asked to wash their hands and then place their right pointer finger on a small lens for approximately 15 seconds. This will be measured immediately following the 3 measured lunch meals at the 3 time points.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure, baseline | Baseline (week 0)
  Systolic and diastolic blood pressure will be measured in duplicate using an automatic monitor fitted with a child-sized cuff. These blood pressure measures will also be converted to sex-, height-, and age-based blood pressure percentiles using an online calculator developed by Baylor College of Medicine. This will be measured on three consecutive days during each of the measurement weeks below.
Systolic and diastolic blood pressure, post-intervention | post-intervention (week 7)
  Systolic and diastolic blood pressure will be measured in duplicate using an automatic monitor fitted with a child-sized cuff. These blood pressure measures will also be converted to sex-, height-, and age-based blood pressure percentiles using an online calculator developed by Baylor College of Medicine. This will be measured on three consecutive days during each of the measurement weeks below.
Systolic and diastolic blood pressure, follow-up | follow-up (week 14)
  Systolic and diastolic blood pressure will be measured in duplicate using an automatic monitor fitted with a child-sized cuff. These blood pressure measures will also be converted to sex-, height-, and age-based blood pressure percentiles using an online calculator developed by Baylor College of Medicine. This will be measured on three consecutive days during each of the measurement weeks below.
Physical activity levels, baseline | Baseline (week 0)
  Physical activity levels will be measured using Actigraph GT3X accelerometers secured with a colorful belt to each child's hip. This data will consist of time spent in the various levels of physical activity (sedentary, light, moderate, and vigorous) and will be measured in 3-day-periods at the time points below. Additionally, parents will be asked to keep a log of when their child is wearing the Actigraph device while at home including the time they take the device off before bed, time they put it on in the morning, and when it is removed for bathing.
Physical activity levels, post-intervention | Post-intervention (week 7)
  Physical activity levels will be measured using Actigraph GT3X accelerometers secured with a colorful belt to each child's hip. This data will consist of time spent in the various levels of physical activity (sedentary, light, moderate, and vigorous) and will be measured in 3-day-periods at the time points below. Additionally, parents will be asked to keep a log of when their child is wearing the Actigraph device while at home including the time they take the device off before bed, time they put it on in the morning, and when it is removed for bathing.
Fruit and vegetable liking, baseline to post-intervention | Change in fruit and vegetable liking from baseline (week 0) to post-intervention (week 7)
  Food liking will be measured during the observed lunch meals using age-appropriate Likert scales that ask children about whether they "like", "neither", or "dislike" the specified food's appearance, smell, taste, and texture, and their overall liking of the food.
Fruit and vegetable liking, baseline to follow-up | Change in fruit and vegetable liking from baseline (week 0) to follow-up (week 14)
  Food liking will be measured during the observed lunch meals using age-appropriate Likert scales that ask children about whether they "like", "neither", or "dislike" the specified food's appearance, smell, taste, and texture, and their overall liking of the food.
Willingness to try fruit and vegetable | Once weekly during the taste-test activity of the nutrition education curriculum (6 weeks total; weeks 1-6)
  Willingness to try foods will be measured during the taste-test activity using the Taste Test Tool that involves asking the children a series of questions including: "Have you ever seen this food before?", "Have you ever tried this food before?", "Did you try this food today?", "Would you try this food again at school?", "Would you try this food again at home?"and "Would you ask for this food at home?" Children will be asked to answer "yes", "no", or "not sure". This will only be measured in the children whose classroom has been allocated to the intervention group (nutrition education curriculum)
Satiety, baseline | Baseline (week 0)
  Satiety will be measured immediately before and after the ad libitum lunch meals where food intake is measured. First, an age-appropriate story will be read to the children to familiarize them with the meanings of "hungry" and "full" and children will be asked to answer questions about the characters' feelings of hunger/fullness based on what they reported eating to ascertain comprehension. Then, satiety will be measured using an age-appropriate 4-point scale developed for preschool children. The children are first asked whether they are hungry or full, and then subsequently asked the intensity of the feeling using "very" or "a little", ie "a little hungry/full" or "very hungry/full".
Satiety, post-intervention | post-intervention (week 7)
  Satiety will be measured immediately before and after the ad libitum lunch meals where food intake is measured. First, an age-appropriate story will be read to the children to familiarize them with the meanings of "hungry" and "full" and children will be asked to answer questions about the characters' feelings of hunger/fullness based on what they reported eating to ascertain comprehension. Then, satiety will be measured using an age-appropriate 4-point scale developed for preschool children. The children are first asked whether they are hungry or full, and then subsequently asked the intensity of the feeling using "very" or "a little", ie "a little hungry/full" or "very hungry/full".
Satiety, follow-up | follow-up (week 14)
  Satiety will be measured immediately before and after the ad libitum lunch meals where food intake is measured. First, an age-appropriate story will be read to the children to familiarize them with the meanings of "hungry" and "full" and children will be asked to answer questions about the characters' feelings of hunger/fullness based on what they reported eating to ascertain comprehension. Then, satiety will be measured using an age-appropriate 4-point scale developed for preschool children. The children are first asked whether they are hungry or full, and then subsequently asked the intensity of the feeling using "very" or "a little", ie "a little hungry/full" or "very hungry/full".
Anthropometrics | Baseline (week 0)
  Each child's height and weight will be measured. This will be used to calculate their BMI-for-age percentile score based on the CDC growth charts.
Food intake during snack, baseline | Baseline (week 0)
  Snack intake (during morning and afternoon snack) will be measured during the same days as the lunch intake measurements, but will use different methods. For snack intake measurements, trained researchers will use visual observation to estimate the children's snack intake that will be recorded using common household measurements (cups, tablespoons, etc). Researchers will each be assigned 4 children to record. They will be asked not to engage with the children. This will be used in their estimate of total energy requirements.
Food intake during snack, post-intervention | Post-intervention (week 7)
  Snack intake (during morning and afternoon snack) will be measured during the same days as the lunch intake measurements, but will use different methods. For snack intake measurements, trained researchers will use visual observation to estimate the children's snack intake that will be recorded using common household measurements (cups, tablespoons, etc). Researchers will each be assigned 4 children to record. They will be asked not to engage with the children. This will be used in their estimate of total energy requirements.
Food intake at home, baseline | Baseline (week 0)
  Parents will be asked to report their child's usual diet using two researcher-conducted, parent-assisted 24-hour dietary recall method. This will occur on the same days that lunch intake and skin carotenoids will be recorded. This will be collected using Nutrition Data System for Research (NDSR) program that has an integrated script for prompting of dietary intake. There are additional supplementary questions following the dietary recall that ask parents to report the amount of time the child spent in sedentary activity and amount of screen time the child engaged in the previous day, both in minutes.
Food intake at home, post-intervention | Post-intervention (week 7)
  Parents will be asked to report their child's usual diet using two researcher-conducted, parent-assisted 24-hour dietary recall method. This will occur on the same days that lunch intake and skin carotenoids will be recorded. This will be collected using Nutrition Data System for Research (NDSR) program that has an integrated script for prompting of dietary intake. There are additional supplementary questions following the dietary recall that ask parents to report the amount of time the child spent in sedentary activity and amount of screen time the child engaged in the previous day, both in minutes.

OTHER OUTCOMES:
Sociodemographic information | Baseline (week 0)
  Parents will be asked to report their own age, race, ethnicity, education level, participation in WIC or SNAP programs, household income and size, and number of children. Parents will be asked to report their child's date of birth, sex, race, ethnicity, allergies, digestive diseases, and developmental delays.
Child eating behavior | Baseline (week 0)
  Parents will be asked to complete a questionnaire that characterizes their child's food neophobia measured using the Food Neophobia scale. Parents will be asked to complete a questionnaire that characterizes their child's eating behavior and relationship with food using a 35-item questionnaire Child Eating Behavior Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Kranz, PhD, Principal Investigator — University of Virginia
Locations (1):
- Westminster Child Care Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be available after publication of results. The name of the childcare centers that participated will not be mentioned in any released data to protect the identity of participating children.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: This data is collected as part of a doctoral dissertation. Data will become available following dissertation defense and publication of results.
Access Criteria: Depends on the journal criteria

REFERENCES:
- [Background] Lioret S, Campbell KJ, McNaughton SA, Cameron AJ, Salmon J, Abbott G, Hesketh KD. Lifestyle Patterns Begin in Early Childhood, Persist and Are Socioeconomically Patterned, Confirming the Importance of Early Life Interventions. Nutrients. 2020 Mar 9;12(3):724. doi: 10.3390/nu12030724. PMID 32182889
- [Background] Livingstone MB, Robson PJ. Measurement of dietary intake in children. Proc Nutr Soc. 2000 May;59(2):279-93. doi: 10.1017/s0029665100000318. PMID 10946797
- [Background] Treiber FA, Leonard SB, Frank G, Musante L, Davis H, Strong WB, Levy M. Dietary assessment instruments for preschool children: reliability of parental responses to the 24-hour recall and a food frequency questionnaire. J Am Diet Assoc. 1990 Jun;90(6):814-20. PMID 2345254
- [Background] Scarmo S, Henebery K, Peracchio H, Cartmel B, Lin H, Ermakov IV, Gellermann W, Bernstein PS, Duffy VB, Mayne ST. Skin carotenoid status measured by resonance Raman spectroscopy as a biomarker of fruit and vegetable intake in preschool children. Eur J Clin Nutr. 2012 May;66(5):555-60. doi: 10.1038/ejcn.2012.31. Epub 2012 Mar 21. PMID 22434053
- [Background] Hodder RK, O'Brien KM, Stacey FG, Wyse RJ, Clinton-McHarg T, Tzelepis F, James EL, Bartlem KM, Nathan NK, Sutherland R, Robson E, Yoong SL, Wolfenden L. Interventions for increasing fruit and vegetable consumption in children aged five years and under. Cochrane Database Syst Rev. 2018 May 17;5(5):CD008552. doi: 10.1002/14651858.CD008552.pub5. PMID 29770960
- [Background] Gripshover SJ, Markman EM. Teaching young children a theory of nutrition: conceptual change and the potential for increased vegetable consumption. Psychol Sci. 2013 Aug;24(8):1541-53. doi: 10.1177/0956797612474827. Epub 2013 Jun 26. PMID 23804961
- [Background] Witt KE, Dunn C. Increasing fruit and vegetable consumption among preschoolers: evaluation of color me healthy. J Nutr Educ Behav. 2012 Mar-Apr;44(2):107-13. doi: 10.1016/j.jneb.2011.01.002. Epub 2011 Sep 16. PMID 21924957
- [Background] Cooke L. The importance of exposure for healthy eating in childhood: a review. J Hum Nutr Diet. 2007 Aug;20(4):294-301. doi: 10.1111/j.1365-277X.2007.00804.x. PMID 17635306
- [Background] Singer MR, Moore LL, Garrahie EJ, Ellison RC. The tracking of nutrient intake in young children: the Framingham Children's Study. Am J Public Health. 1995 Dec;85(12):1673-7. doi: 10.2105/ajph.85.12.1673. PMID 7503343
- [Background] Wuhl E. Hypertension in childhood obesity. Acta Paediatr. 2019 Jan;108(1):37-43. doi: 10.1111/apa.14551. Epub 2018 Sep 19. PMID 30144170
- [Background] Miguel-Berges ML, Zachari K, Santaliestra-Pasias AM, Mouratidou T, Androutsos O, Iotova V, Galcheva S, De Craemer M, Cardon G, Koletzko B, Kulaga Z, Manios Y, Moreno LA. Clustering of energy balance-related behaviours and parental education in European preschool children: the ToyBox study. Br J Nutr. 2017 Dec;118(12):1089-1096. doi: 10.1017/S0007114517003129. Epub 2017 Dec 4. PMID 29198192
- [Background] Kranz S, Brauchla M, Campbell WW, Mattes RD, Schwichtenberg AJ. High-Protein and High-Dietary Fiber Breakfasts Result in Equal Feelings of Fullness and Better Diet Quality in Low-Income Preschoolers Compared with Their Usual Breakfast. J Nutr. 2017 Mar;147(3):445-452. doi: 10.3945/jn.116.234153. Epub 2017 Jan 11. PMID 28077732